CLINICAL TRIAL: NCT04423575
Title: Clinical and Economic Evaluation of Outpatient Bariatric Surgery
Brief Title: Outpatient Bariatric Surgery
Acronym: Bariatric Ambu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-011
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Morbid
Keywords: Severe Obesity; Outpatient Surgery; Bariatric Surgery; Roux-en-Y Gastric Bypass; Sleeve Gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatients (Experimental): Health care pathway: patient education, communication to liberal nurses, first-position surgical planning, bariatric surgery (bypass or sleeve) as outpatient procedure, follow-up by home nurse twice-a-day, standardized communication to surgeons, management of possible complications
  Interventions: Other: Outpatient health care pathway
- Inpatients (No Intervention): Standard care pathway with bariatric surgery (bypass or sleeve) as inpatient procedure (at least one night in the hospital)

INTERVENTIONS:
Other: Outpatient health care pathway — A surgical procedure performed as an outpatient procedure means that the patient leaves the hospital before 8pm the same day. The surgery is identical but the standard care pathway is reinforced to insure a safe return to home.
  Arms: Outpatients

SUMMARY:
This study first presents the organizational path and the health interventions included in the care episode for outpatient bariatric surgery, as compared to the health interventions usually performed in the care episode for bariatric surgery (including a conventional hospitalization with at least one-night inpatient). Then, the study aims to estimate and to compare the costs of bariatric surgery inpatient care episode to the costs of outpatient care episode, and also to evaluate the postoperative medical consequences.

DETAILED DESCRIPTION:
This study first presents the organizational path and the health interventions included in the care episode for outpatient bariatric surgery, as compared to the health interventions usually performed in the care episode for bariatric surgery (including a conventional hospitalization with at least one-night inpatient).

This single-center, matched case-control study will be conducted in the Endocrine and Digestive Surgery Unit, Center of Excellence in Bariatric Surgery, of the University Hospital of Strasbourg. All the patients scheduled for bariatric procedures (Roux-en-Y gastric bypass and Sleeve Gastrectomy) and eligible for outpatient ambulatory procedures, will be checked for the inclusion criteria and will be asked if they accepted the outpatient bariatric procedure. If they accept, they will be included in the group A ("Outpatients"). At the end of the inclusion period, the patients in group A will be paired to patients who were operated in the same period, who had a conventional hospitalization and who will be matched based on the type of intervention, the age and the ASA status. These patients will form the group B ("Inpatients").

The integrated care pathway of the outpatients was formalized in order to secure this care pathway. It includes: patient education, enhanced rehabilitation program, first-position surgical planning, follow-up by home nurse twice-a-day, standardized communication to surgeons, and management of possible complications. All the health care interventions (anticipated or not) will be recorded for both groups.

The study aims to estimate and to compare the costs of bariatric surgery inpatient care episode to the costs of outpatient care episode, and also to evaluate the postoperative medical consequences. A cost-minimization analysis will be performed from the perspective of the healthcare provider. The direct costs of care production will be considered and estimated by a micro-costing methodology. The time horizon is set from the pre-operative outpatient appointment with the bariatric surgeon to the one-month post-operative appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patient between the age of 18 and 60
* Patient with a BMI of more than 35 with comorbidities or BMI of more than 40
* Speaking and understanding French
* Access to a phone
* Access to a suitable healthcare facility near his residence
* Appropriate post-operative residence
* Moderate and/or controlled comorbidities
* Patient able to understand research objectives and risks and to give informed consent
* Patient not living alone
* affiliated to the French health insurance system

Exclusion Criteria:

* patient unable to provide informed consent
* Previous bariatric surgery
* Previous laparotomy
* BMI of more than 50
* Insulin-dependent diabetes
* Uncorrected preoperative anaemia
* Anticoagulation that cannot be interrupted
* Ischemic heart disease
* Untreated obstructive sleep apnea syndrome (OSA)
* dialysis
* Liver cirrhosis
* Subject under guardianship, curatorship, safeguarding/protection of justice
* Pregnancy
* Breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Mean cost evaluation of health care pathway | from the pre-operative appointment with the bariatric surgeon to the one-month post-operative appointment
  Mean costs related to the described health care pathway (outpatients vs inpatients) will be assessed by micro-costing methodology

SECONDARY OUTCOMES:
Mean hospital length of stay | from surgery to one month postoperatively
  Mean hospital length of stay including readmission duration
Quality of life evaluation: EQ-5D (EuroQoL-5 Dimensions) scale | at day 0, day 7 and day 30 postoperatively
  The EQ-5D Quality of Life scale consists of :
  (i) a descriptive system, consists in 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
  (ii) a visual analog scale, records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state" and "Worst imaginable health state".
Complication rate | from surgery to one month postoperatively
  rate of postoperative complications
Ambulatory failure rate | from surgery to one month postoperatively
  rate of patients in Arm 1 who spent at least the first night in the hospital
Readmission rate | from surgery to one month postoperatively
  rate of patients in Arm 1 who were readmitted in the hospital, after being successful dismissed at day 0
Costs related to Complication | from surgery to one month postoperatively
  costs related to the postoperative complications will be assessed by micro-costing methodology

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela IGNAT, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg
Locations (1):
- University Hospital of Strasbourg, Department of Digestive and Endocrine Surgery, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cobourn C, Mumford D, Chapman MA, Wells L. Laparoscopic gastric banding is safe in outpatient surgical centers. Obes Surg. 2010 Apr;20(4):415-22. doi: 10.1007/s11695-009-0065-7. PMID 20077029
- [Background] McCarty TM, Arnold DT, Lamont JP, Fisher TL, Kuhn JA. Optimizing outcomes in bariatric surgery: outpatient laparoscopic gastric bypass. Ann Surg. 2005 Oct;242(4):494-8; discussion 498-501. doi: 10.1097/01.sla.0000183354.66073.4c. PMID 16192809
- [Background] Ignat M, Vix M, Imad I, D'Urso A, Perretta S, Marescaux J, Mutter D. Randomized trial of Roux-en-Y gastric bypass versus sleeve gastrectomy in achieving excess weight loss. Br J Surg. 2017 Feb;104(3):248-256. doi: 10.1002/bjs.10400. Epub 2016 Nov 30. PMID 27901287
- [Derived] Ignat M, Ansiaux J, Osailan S, D'Urso A, Morainvillers-Sigwalt L, Vix M, Mutter D. A Cost Analysis of Healthcare Episodes Including Day-Case Bariatric Surgery (Roux-en-Y Gastric Bypass and Sleeve Gastrectomy) Versus Inpatient Surgery. Obes Surg. 2022 Aug;32(8):2504-2511. doi: 10.1007/s11695-022-06144-3. Epub 2022 Jun 10. PMID 35689142
- See also: Epidemiologic study on obesity in France, 2017 — https://www.santepubliquefrance.fr/determinants-de-sante/nutrition-et-activite-physique/documents/rapport-synthese/etude-de-sante-sur-l-environnement-la-biosurveillance-l-activite-physique-et-la-nutrition-esteban-2014-2016.-volet-nutrition.-chapitre-corpulence
- See also: Epidemiologic study on obesity surgery in France, 2018 — http://beh.santepubliquefrance.fr/beh/2018/5/pdf/2018_5_3.pdf